CLINICAL TRIAL: NCT03326427
Title: Randomized Clinical Trial With Adapted Skill Training Group From Dialectical Behavior Therapy as add-on Treatment for Adults With Attention Deficit/Hyperactive Using Medication
Brief Title: Group Dialectical Behavior Therapy as add-on Treatment for Adults With Attention Deficit/Hyperactive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0358; 65041316400005327 (Other: CAAE)
Record Dates: First submitted 2017-10-09; First posted 2017-10-31 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactive Disorder; Skill Training Group; Dialectical Behavior Therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skill Training Group (Experimental): A twelve sessions protocol of the Skill Training Group of the Dialectical Behavior Therapy.
  Interventions: Behavioral: Skill Training Group of the Dialectical Behavior Therapy
- Treatment as Usual (Active Comparator): Patients will have one psychiatric session to control their medication adherence.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Skill Training Group of the Dialectical Behavior Therapy — A 12 session version of the Skill Training Group of the Dialectical Behavior Therapy, adapted for treatment of ADHD.
  Arms: Skill Training Group
Other: Treatment as Usual — Conventional protocol using only medication (including drug adherence).
  Other Names: waiting list
  Arms: Treatment as Usual

SUMMARY:
Attention-Deficit/Hyperactive Disorder (ADHD) in adults is associated with global impairments and deficits in quality of life. The ADHD functional impairments during adulthood usually persist even after adequate medication treatment. The Skill Training Group of the Dialectical Behavioral Therapy (DBT) is one of the group therapies that had been adapted for the specific treatment of ADHD patients. Our primary aim is to explore the feasibility of the approach in different culture and to evaluate the efficacy of the Skill Training Group as an add-on treatment for adults using ADHD medication. This is a Randomized Clinical Trial comparing the Skill Training Group added to stimulants to treatment as usual. 52 adults previously diagnosed with ADHD and treated with stimulants in our ADHD outpatient program will be enrolled. Only patients with residual symptoms will be included (ADHD-Self Report Scale - ASRS ≥ 20). The intervention comprises the standard 12 sessions therapy program. The groups will have between 8 and 12 patients each, and will be conducted by a trained DBT therapist with supervision from a senior DBT therapist. The primary outcome will be the ASRS scores. Secondary outcomes include scores in ADHD Quality of Life, Beck's Depression Inventory, Beck's Anxiety Inventory, and performance in a neuropsychological test (difference between pre and post-intervention) (Stop Signal Task). Adherence to the protocol will also be checked. The recruitment was initially scheduled for beginning in November.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADHD
* Medicated with following drugs and minimum daily dosages:

Methylphenidate ≥ 0.5 mg/kg Lisdexamfetamine ≥ 30mg Bupropion ≥ 150 mg Modafinil ≥ 200mg Imipramine ≥ 1mg/kg

* At least one month of stabilized dosage for any psychiatric medication.
* ADHD-Self Report Scale ≥ 20.
* Knowledge of oral and written communication in Portuguese
* IQ>85 (intelligence quotient)

Exclusion Criteria:

* diagnoses of Borderline or Anti-social personality disorders.
* diagnoses of autism spectrum disorder
* current episode of major depression or suicide toughs
* current episodes of mania or hypomania
* recent episodes of drug abuse (last 6 months)
* diagnoses of drug dependence
* patients that change their medications or their psychiatric conditions in the exclusion criteria above after the beginning of the protocol will have their data censored, but included in the intention to treat analyses. These patients will keep the right to attend all the sessions in the protocol at their discretion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2018-11-24 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Change in Adult Attention-Deficit/Hyperactive Disorder Self Rating Scale | 12 Weeks
  Sefl rated scale to measure Attention Deficit Hyperactive Disorder Symptoms Symptoms.
  ASRS has 18 questions about ADHD symptoms. Each question is scored between 0 (never happen), and 4 (very frequently). The total score goes from 0 up to 72. Higher scores mean more symptoms and higher ADHD's impairments.

SECONDARY OUTCOMES:
Change in Attention-Deficit/Hyperactive Disorder Self Rating Scale - Mid-treatment | 6 Weeks
  Sefl rated scale to measure Attention Deficit Hyperactive Disorder Symptoms. ASRS has 18 questions about ADHD symptoms. Each question is scored between 0 (never happen), and 4 (very frequently). The total score goes from 0 up to 72. Higher scores mean more symptoms and higher ADHD's impairments.
Change in Attention-Deficit/Hyperactive Disorder Quality of Life | 12 Weeks
  "Adult Attention-Deficit/Hyperactivity Disorder Quality-of-Life Scale (AAQoL)" is a Self-rated scale for quality of life in ADHD.
  The scale has 29 questions ranging from 1 to 5. The AaQol focuses on four areas of patients quality of life: mental health, life goals, productivity, and relationships. The total scores go from 0 to 145. Higher scores mean the patient has a worse perception of his quality of life.
Change in Attention-Deficit/Hyperactive Disorder Quality of Life - Mid-treatment | 6 weeks
  "Adult Attention-Deficit/Hyperactivity Disorder Quality-of-Life Scale (AAQoL)" is a Self-rated scale for quality of life in ADHD.
  The scale has 29 questions ranging from 1 to 5. The AaQol focuses on four areas of patients quality of life: mental health, life goals, productivity, and relationships. The total scores go from 0 to 145. Higher scores mean the patient has a worse perception of his quality of life.
Change in Beck Depression Inventory | 12 Weeks
  Beck Depression Inventory (BDI) is a Self-rated scale for depression. BDI has 21 questions ranging from 0-4, with the maximum score being 63. Higher scores mean higher depression levels. Scores between 0-13 are considered minimal depression, between 14 and 19 are considered mild depression, from 20 to 28 moderate depression, over 29 are considered severe depression.
Change in Beck Depression Inventory - Mid-treatment | 6 Weeks
  Beck Depression Inventory (BDI) is a Self-rated scale for depression BDI has 21 questions ranging from 0-4, with the maximum score being 63. Higher scores mean higher depression levels. Scores between 0-13 are considered minimal depression, between 14 and 19 are considered mild depression, from 20 to 28 moderate depression, over 29 are considered severe depression.
Change in Beck Anxiety Inventory | 12 Weeks
  Beck Anxiety Inventory is a Self-rated scale for anxiety. BAI has 21 questions ranging from 0-4, with the maximum score being 63. Higher scores mean higher anxiety levels. Scores between 0-9 are considered normal, between 10 and 18 are considered mild to moderate anxiety, from 19 to 29 moderate to severe anxiety, over 30 are considered severe anxiety.
Change in Beck Anxiety Inventory - Mid-treatment | 6 Weeks
  Beck Anxiety Inventory is a Self-rated scale for anxiety. BAI has 21 questions ranging from 0-4, with the maximum score being 63. Higher scores mean higher anxiety levels. Scores between 0-9 are considered normal, between 10 and 18 are considered mild to moderate anxiety, from 19 to 29 moderate to severe anxiety, over 30 are considered severe anxiety.
Change in the reflexive function questionnaire | 12 weeks
  A self-reported scale to measure reflexive psychological functions. The questionnaire has 8 questions variating from one to seven. Total scores have ranged between 8 and 56. Better reflexive functions mean lowers scores on the scale.
Change in the reflexive function questionnaire - Mid-treatment | 6 weeks
  A self-reported scale to measure reflexive psychological functions. The questionnaire has 8 questions variating from one to seven. Total scores have ranged between 8 and 56. Better reflexive functions mean lowers scores on the scale.
Change in the Go NoGo | 14 weeks
  Computer-based psychometric task. Consists of three stimuli, one green arrow to left, one pointing to the right, and one arrow pointing to both sides. Subjects have to press correctly to right or left in the presence of the correspondent arrow or do not press any in the presence of the arrow to both sides. The task takes around 5 minutes.
  The aim is to measure impulsivity through response times, commissions and errors.
Change in Stroop Task | 14 Weeks
  neuropsychological test to measure response inhibition (impulse control). The task has four stimuli, two green arrows, pointing to the right or left, and two red arrows, pointing to the right or left. When the green stimuli appear the subject must press the button to the correspondent side, in the appearance of the red stimuli the subject must press a button of the opposing side.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Augusto Rohde, Principal Investigator — UNIVERSIDADE FEDERAL DO RIO GRANDE DO SUL (UFRGS)
Locations (1):
- Centro de Pesquisa Clínica, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
Patient's individual data will be available only for the researchers and additional members of the research team, and for the patients it self.

REFERENCES:
- [Derived] Moritz GR, Pizutti LT, Cancian ACM, Dillenburg MS, de Souza LAS, Lewgoy LB, Basso P, Andreola MMP, Bau CHD, Victor MM, Teche SP, Grevet EH, Philipsen A, Rohde LAP. Feasibility trial of the dialectical behavior therapy skills training group as add-on treatment for adults with attention-deficit/hyperactivity disorder. J Clin Psychol. 2021 Mar;77(3):516-524. doi: 10.1002/jclp.23049. Epub 2020 Sep 2. PMID 32880953
- See also: The therapy protocol that will be used at the research — https://www.ncbi.nlm.nih.gov/pubmed/26536057